CLINICAL TRIAL: NCT02680444
Title: Exploring Daily Affective Changes in University Students With a Mindful Positive Reappraisal Intervention: a Daily Diary Randomized Controlled Trial
Brief Title: Mindful Positive Reappraisal: a Daily Diary Randomized Controlled Trial
Acronym: Reappraisal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekaterina Pogrebtsova (Other)
Responsible Party: Sponsor-Investigator, Ekaterina Pogrebtsova, Graduate Researcher, University of Guelph
Organization: University of Guelph (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 11NV038
Record Dates: First submitted 2016-02-04; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Mental Health Wellness 1
Keywords: Mindfulness; Primary Promotion; Mental Health; Well-being; Positive Reappraisal
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reappraisal-Only Intervention (Experimental): Participants were instructed to independently practice the Self-Administered Reappraisal-Only Exercise in the evening for five days. First, participants recalled a negative event from that day and then followed the positive reappraisal instructions available online. This involved thinking about how one could grow, learn or benefit from the negative event in any way possible.
  Interventions: Behavioral: Self-Administered Reappraisal-Only Exercise
- Mindful-Reappraisal Intervention (Experimental): Participants were instructed to independently practice the Self-Administered Mindful-Reappraisal Exercise in the evening for five days. First, participants recalled a negative event from that day and then followed the Mindful-Reappraisal instructions available online. This involved thinking about the negative event in an objective, non-judgmental way, then following the Reappraisal-Only instructions, and closing off with a brief mindfulness breathing technique.
  Interventions: Behavioral: Self-Administered Mindful-Reappraisal Exercise
- Event Recall Active Control (Active Comparator): Participants were instructed to independently practice the Self-Administered Event Recall Exercise in the evening for five days. In this condition, participants were only instructed to recall a negative event from that day with no reappraisal exercise.
  Interventions: Behavioral: Self-Administered Event Recall Exercise

INTERVENTIONS:
Behavioral: Self-Administered Mindful-Reappraisal Exercise — Combining the practice of mindful acceptance of negative events combined with a reappraisal of the event by examining its positive aspects.
  Arms: Mindful-Reappraisal Intervention
Behavioral: Self-Administered Reappraisal-Only Exercise — A reappraisal of daily negative events by examining the positive aspects.
  Arms: Reappraisal-Only Intervention
Behavioral: Self-Administered Event Recall Exercise — Recall a negative event that took place that day.
  Arms: Event Recall Active Control

SUMMARY:
Brief and cost-effective interventions teaching emotion regulation techniques can be feasibly applied to promote mental health in University students. The tools of mindfulness (i.e., objective awareness and acceptance) and positive reappraisal (i.e., positive re-evaluation of negative events) can mutually benefit one another to promote well-being. The current study explored the effects of a randomly-assigned Mindful-Reappraisal intervention (n=36) compared to Reappraisal-Only (n=34) and an active control (n=36) on university students' daily affect over five days. Time by condition interactions were analyzed with planned contrasts and multilevel growth modelling.

DETAILED DESCRIPTION:
The University student lifestyle can lead to heightened stress, anxiety, and burnout. To promote mental health, brief and cost-effective interventions teaching beneficial emotion regulation techniques can not only counteract the negative but also foster positive functioning. The tools of mindfulness (i.e., objective awareness and acceptance) and positive reappraisal (i.e., positive re-evaluation of negative events) can mutually benefit one another to promote well-being. However, there is currently little research testing the viability of brief, self-administered interventions combining training of mindfulness and positive reappraisal. The current study explored the effects of a randomly-assigned Mindful-Reappraisal intervention (n=36) compared to Reappraisal-Only (n=34) and an active control (n=36) on university students' daily affect over five days. Time by condition interactions were analyzed with planned contrasts and multilevel growth modelling.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students

Exclusion Criteria:

* Not undergraduate students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Daily Affect | Day 1 - Day 5 of the intervention practice days
  Daily affect was measured with two scales (i.e., positive affect and negative affect) and assessed participants' general affect over the past 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: M. Gloria Gonzalez-Morales, Principal Investigator — University of Guelph

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available.